CLINICAL TRIAL: NCT01748461
Title: Objective Assessment and Promotion of Physical Activity in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: ML8733
Record Dates: First submitted 2012-12-03; First posted 2012-12-12 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Elderly
Keywords: intervention study in elderly (65+); cycle ergometer; physical activity; physical fitness; assisted living facility
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Structured intervention (Active Comparator): Supervised cycle ergometer program
  Interventions: Behavioral: Structured intervention
- Coach intervention (Active Comparator): Non-supervised cycle ergometer program
  Interventions: Behavioral: Coach intervention
- Control group (No Intervention): No cycle ergometer program

INTERVENTIONS:
Behavioral: Structured intervention — 3x/week - 10 weeks - Support by fitness instructor - Individualised exercise program (cycle ergometer)
  Arms: Structured intervention
Behavioral: Coach intervention — promote autonomy - 4 visits during 10 weeks - Support by coach (encouragement) - Individualised exercise program
  Arms: Coach intervention

SUMMARY:
The purpose of the present study is to evaluate the short-term and long-term effects of a cycle ergometer program on physical activity and physical fitness in elderly (65+). Therefore, physical activity, physical fitness and functionality are measured at baseline, after 10 weeks (after the intervention period), after 6 months and after 1 year.

Different coaching techniques (to promote the use of a cycle ergometer and cycle ergometer program) will also be evaluated. What is the best (coaching) approach for long-term adherence (physical activity)?

ELIGIBILITY:
Inclusion Criteria:

* 65 yrs
* residents of a service flat
* No frequent use of bike / cycle ergometer

Exclusion Criteria:

* recent cardiovascular event or fracture
* vestibular or thrombotic disorder
* severe dementia
* need for oxygen supplementation during daily activities

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 105 (Actual)
Dates: Start 2013-05; Primary Completion 2014-01 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change in objective and subjective measures of degree of physical activity | baseline, 10 weeks, 6 months, 1 year
  Physical activity will be measured using a standardized questionnaire and a Sensewear. A Sensewear is an activity monitor (accelerometer) carried on the upper arm during several days and registers the amount of physical activity.
Change in objective measures of physical fitness | baseline, 10 weeks, 6 months, 1 year
  Physical fitness will be measured using a standardized Six-Minute Walk Test and a Six-Minute Cycle Test.
Change in objective measures of functionality | baseline, 10 weeks, 6 months, 1 year
  Functionality will be measured using the standardized The Physical Performance Test and 2 strength tests (hand grip and knee extension).

SECONDARY OUTCOMES:
Change in mental well-being | baseline, 10 weeks, 6 months, 1 year
  Standardized questionnaire
Change in motivation to be physically active | baseline, 10 weeks, 6 months, 1 year
  Standardized questionnaire
Change in self-efficacy to be physically active | baseline, 10 weeks, 6 months, 1 year
  Standardized questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Kinesiology and Rehabilitation Sciences, Leuven, Belgium